CLINICAL TRIAL: NCT03646526
Title: Bioavailability Study of Amitriptyline Hydrochloride Tablets
Acronym: AMTL-BE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Hunan DongtingPharm.Co.Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ZYYY-AMTL-BE-2018-02
Record Dates: First submitted 2018-05-18; First posted 2018-08-24 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-01

CONDITIONS: Depressive Disorder
Keywords: Amitriptyline hydrochloride
MeSH Terms: conditions — Depressive Disorder | interventions — Amitriptyline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fast group (Experimental): During the study session, healthy subjects will be administered a single dose of Amitriptyline Hydrochloride 25Mg Tablet（Hunan Dongting） or Amitriptyline Hydrochloride 25Mg Tablet（Sandoz） under fasting condition .
  cycle 1 Drug: Amitriptyline Hydrochloride 25Mg Tablet（Hunan Dongting）/cycle 2 Drug: Amitriptyline Hydrochloride 25Mg Tablet（Sandoz） or cycle 1 Drug: Amitriptyline Hydrochloride 25Mg Tablet（Sandoz）/cycle 2 Drug: Amitriptyline Hydrochloride 25Mg Tablet（Hunan Dongting）
  Interventions: Drug: Amitriptyline Hydrochloride 25Mg Tablet（Hunan Dongting）; Drug: Amitriptyline Hydrochloride 25Mg Tablet（Sandoz）
- Feeding group (Experimental): During the study session, healthy subjects will be administered a single dose of Amitriptyline Hydrochloride 25Mg Tablet（Hunan Dongting） or Amitriptyline Hydrochloride 25Mg Tablet（Sandoz） under feeding condition.
  cycle 1 Drug: Amitriptyline Hydrochloride 25Mg Tablet（Hunan Dongting）/cycle 2 Drug: Amitriptyline Hydrochloride 25Mg Tablet（Sandoz） or cycle 1 Drug: Amitriptyline Hydrochloride 25Mg Tablet（Sandoz）/cycle 2 Drug: Amitriptyline Hydrochloride 25Mg Tablet（Hunan Dongting）
  Interventions: Drug: Amitriptyline Hydrochloride 25Mg Tablet（Hunan Dongting）; Drug: Amitriptyline Hydrochloride 25Mg Tablet（Sandoz）

INTERVENTIONS:
Drug: Amitriptyline Hydrochloride 25Mg Tablet（Hunan Dongting） — Amitriptyline Hydrochloride 25Mg Tablet（Hunan Dongting）is a generic product manufactured by Hunan Dongting Pharmaceutical Co., Ltd.
Drug: Amitriptyline Hydrochloride 25Mg Tablet（Sandoz） — Amitriptyline Hydrochloride 25Mg Tablet（Sandoz）is a generic product manufactured by Sandoz Inc;

SUMMARY:
Main Objectives: In Chinese healthy subjects under both fasting and postprandial conditions, amitriptyline hydrochloride tablets (size: 25 mg) produced by Sandoz Inc., US Orange Book, were used as reference preparations. A single-dose oral reference preparation and amitriptyline hydrochloride tablets (size: 25 mg) produced by Hunan Dongting Pharmaceutical Co., Ltd., and the calculation of the drug by the time course of amitriptyline and its active metabolite, nortriptyline, in vivo The kinetic parameters were compared, and the relative bioavailability of the two was compared to evaluate bioequivalence, which provided the basis for the bioequivalence study of amitriptyline hydrochloride tablets by Hunan Dongting Pharmaceutical Co., Ltd.

Secondary Objective: To monitor the safety of fasting and postprandial oral test and reference preparations.

DETAILED DESCRIPTION:
This clinical study is a single-center, randomized, open clinical study divided into two parts, the first part is the pre-test and the second part is the formal test.

Both pre-test and formal trials were designed using two preparations, two cycles, and a self-crossover controlled trial.

Twelve subjects were enrolled in the pre-test and randomly divided into two groups. Each group received 25 mg of the test preparation or reference preparation in the first day of each cycle, before the administration (0 h) and after the administration 0.5 h, 1.0 h, 2.0 h, 2.5 h, 3.0 h, 3.5 h, 4.0 h, 4.5 h, 5.0 h, 5.5 h, 6.0 h, 7.0 h, 8.0 h, 10.0 h, 12.0 h, 24.0 h, 36.0 h, 48.0 h, 72.0 h, 96.0 h, 120.0 h, 144 h, 168 h, and 192 h blood samples were measured for plasma amitriptyline concentration for bioequivalence analysis, and the concentration of the active metabolite nortriptyline was determined as supportive evidence of comparable efficacy. The pre-test results will provide the basis for formal testing. The cleaning period is 21 ± 1 day.

The formal trials were divided into fasting and postprandial trials to evaluate the bioequivalence of the test preparation and the reference preparation in a single dose of hollow and postprandial administration in healthy Chinese subjects. Fasting and postprandial trials were enrolled in 24 subjects and randomly divided into 2 groups. Each group received 25 mg of the test preparation or reference preparation on the first day of each cycle, before the administration (0 h) and after the administration 0.5 h, 1.0 h, 2.0 h, 3.0 h, 4.0 h, 5.0 h, 6.0 h, 7.0 h, 8.0 h, 10.0 h, 12.0 h, 24.0 h, 36.0 h, 48.0 h, 72.0 h, 96.0 h, 120.0 h and 144 h blood samples were measured for plasma concentrations of amitriptyline for bioequivalence analysis， and the concentration of the active metabolite nortriptyline was determined as supportive evidence of comparable efficacy.. The cleaning period is 21 ± 1 day.

Based on the results of the first part of the pre-test evaluation, the experimental design and sampling time and other contents of the second part of the formal test may require necessary modifications.

The fasting test and the postprandial test in the formal test were carried out independently.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-45 years old (including 18 and 45 years old), both male and female;
2. Male subjects weigh more than 50kg (including 50kg) and female subjects weigh more than 45kg (including 45kg); Body mass index [BMI = body weight (kg)/height (m)2] is in the range of 19 to 26 kg/m2;
3. According to past medical history, comprehensive physical examination and prescribed laboratory tests, the investigator determined that Healthy subjects;
4. Women of childbearing age have a negative blood pregnancy test and are effective from 14 days before dosing to 6 months after the end of study Appropriate contraceptive measures;
5. Male volunteers must take effective and appropriate 14 days before dosing until 6 months after the end of the study.

   The contraceptive measures and agrees not to perform sperm donation within six months from the administration until the end of the study;
6. Fully understand the purpose of the test, the nature of the test, the study procedures, and possible adverse reactions.

   Willing to participate in the trial and sign the informed consent form (the process of obtaining the informed consent accords with GCP regulations);
7. Communicate well with the researcher, follow the requirements of the entire study, and be willing to stay in the Phase I clinical research ward as required.

Exclusion Criteria:

1. Can not tolerate venipuncture, who have a history of dizziness and pinching blood;
2. Clearly have a history of allergies to the drug ingredients or similar species or to two or more other drugs Sensitive history and highly sensitive to food and environmental substances;
3. Have a history of any serious clinical illness, including but not limited to digestive system, cardiovascular system, respiratory system, Urinary system, musculoskeletal system, endocrine system, neuropsychiatric system, blood system, immune system Patients with a history of diseases and metabolic disorders;
4. Laboratory tests (blood routine, urine routine, blood chemistry, etc.) and chest X-ray and ECG within 2 weeks before the test Those who have abnormal clinical findings
5. Hematological screening (HIV antibody or HBV surface antigen or HCV antibody or TP antibody) positive;
6. women who are breastfeeding, pregnant or plan to become pregnant recently;
7. Female subjects are in lactation or positive pregnancy test during the screening period or during the trial;
8. Male and female subjects who have not taken effective contraception or whose spouse plans to have children within six months;
9. Persons with mental or legal disabilities;
10. Screening for history of prescription drug abuse and/or history of illegal drug abuse within the first 6 months of screening;
11. A person who has a history of alcohol abuse within the first 6 months of screening, ie drinking more than 14 units of alcohol per week (1 unit = 12 ounces or 360 mL beer, 1.5 ounces or 45 mL alcohol 40% spirits, 5 ounces or 150mL wine);
12. Smoke more than 5 cigarettes per day within 6 months before screening;
13. positive for substance abuse screening or alcohol testing;
14. Those with a history of hospitalization or surgery within 3 months prior to screening (excluding appendicitis);
15. Participate in other drug clinical trials within 3 months before screening;
16. Have blood donation or acute blood loss history (≥400 mL) within the first 2 months of screening or 1 after the end of the trial Intended to donate blood during the month;
17. Those who used any other medicine within 2 weeks before the test (prescription drugs, non-prescription drugs, any vitamins) Products or herbs);
18. Drink more than 1L of tea, coffee, and/or caffeinated beverages daily;
19. Those who have special dietary requirements and cannot accept a unified diet;
20. Those who are lactose intolerant (have been drinking milk diarrhea);
21. Those who do not understand the content of the informed consent and those who do not meet the criteria for the trial enrollment;
22. Subjects are poorly adhered to, or the investigator believes there are any individuals who are unfit to participate in the trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Cmax | 144 hours post-dose on Day 1,22
  Maximum Observed Plasma Concentration for amitriptyline
Tmax | 144 hours post-dose on Day 1,22
  Time to Reach the Maximum Plasma Concentration
AUC(0-inf) | 144 hours post-dose on Day 1,22
  Area Under the Plasma Concentration-time Curve from Time 0 to Infinity for amitriptyline
AUC(0-144h) | 144 hours post-dose on Day 1,22
  Area Under the Plasma Concentration-Time Curve From Time 0 to 36 hours Postdose for amitriptyline

CONTACTS AND LOCATIONS:
Overall Officials: Jian LIU, Master, Study Chair — The First Affiliated Hospital,ZheJiang Univercity
Locations (1):
- The First Affiliated Hospital,ZheJiang Univercity, Hanzhou, Zhejiang, China

REFERENCES:
- [Derived] Zhai Y, Wu L, Zheng Y, Wu M, Huang Y, Huang Q, Shentu J, Zhao Q, Liu J. Bioequivalence Study of Amitriptyline Hydrochloride Tablets in Healthy Chinese Volunteers Under Fasting and Fed Conditions. Drug Des Devel Ther. 2020 Aug 4;14:3131-3142. doi: 10.2147/DDDT.S258173. eCollection 2020. PMID 32801649